CLINICAL TRIAL: NCT01306838
Title: Early Supplementation of Enteral Lipid With Combination of Microlipid and Fish Oil in Infants With Enterostomy
Brief Title: Early Provision of Enteral Microlipid and Fish Oil to Infants With Enterostomy
Acronym: EMLFO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00011501
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Short Bowel Syndrome; Necrotizing Enterocolitis; Small Intestine Perforation
Keywords: Short bowel syndrome; Necrotizing enterocolitis; Small intestine perforation; Enterostomy; Intralipid; Microlipid; Fish oil
MeSH Terms: conditions — Short Bowel Syndrome; Enterocolitis, Necrotizing | interventions — Safflower Oil; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The treatment arm is given early enteral supplementation with MicroLipid and Fish oil.
  Interventions: Dietary Supplement: MicroLipid and fish oil
- Control Group (Active Comparator): Routine care
  Interventions: Other: Routine care

INTERVENTIONS:
Dietary Supplement: MicroLipid and fish oil — Infants in treatment arm will receive the same nutrition support as control group before they tolerate enteral feeding at 20 ml/kg/day. Then they will receive study oils when feeds reach 30 ml/kg/day.
  Arms: Treatment
Other: Routine care — Routine care
  Arms: Control Group

SUMMARY:
Necrotizing enterocolitis (NEC) and intestinal perforation are common in premature infants. Often surgery is needed to remove the dead bowel and create an ostomy (a temporary intestinal opening on the infant's abdomen). Infants with ostomies cannot digest and absorb food well, and must receive nutrition through the blood stream, i.e. parental nutrition (PN). However, prolonged dependence on PN can severely damage the liver and gut. Therefore, giving nutrition through the gut, i.e. enteral nutrition, is the primary treatment for infants with ostomies.

Enteral fats, especially polyunsaturated fatty acids (PUFA), are most beneficial in stimulating gut mucosal adaptation, which begins 24 to 48 hours following bowel resection. In addition, the premature intestine has a rapid growth rate. It is likely that the current clinical practice of giving a relatively low-fat diet to infants with ostomies may not meet their high metabolic needs.

The investigators hypothesize that increasing dietary fat content by early supplementation with MicroLipid® (ML, n-6 PUFA) and fish oil (FO, n-3 PUFA) to preserve the proper balance of n-6 and n-3 PUFA, may (i) improve bowel adaptation and infant growth; (ii) reduce the use of PN; and (iii) prevent liver damage and/or cholestasis (jaundice) in infants with ostomies.

DETAILED DESCRIPTION:
It is an interventional randomized open-labeled controlled trial with two groups:

Treatment group: early supplementation of enteral lipid with ML and FO; Control group: routine care.

The primary goal of this study is to obtain pilot data that will inform the subsequent design and execution of a large, randomized trial which will test the hypothesis that infants with short bowel syndrome or ostomy will experience beneficial growth effects from enteral nutrition supplemented with balanced n6/n-3 PUFA, a simple, inexpensive and noninvasive intervention. This pilot study will confirm the safety of PUFA supplemented enteral nutrition, establish the length and amount of enteral versus parenteral nutrition required, and determine the impact on infant growth and intestinal adaptation by measuring expression of four key genes that play a crucial role in intestinal adaptation.

ELIGIBILITY:
Inclusion Criteria:

* infants (age range: newborn to 2-month-old) who are admitted to BCH NICU with a jejunostomy or ileostomy (from surgical intervention for NEC, bowel perforation, midgut volvulus (twisted bowel), atresia or other gastrointestinal surgery);
* who are expected to need full or partial PN for at least 21days from the day of enterostomy placement; and
* have received enteral feedings ≤ 4 days since enterostomy placement

Exclusion Criteria:

* infant with colostomy;
* infants with enterostomy but

  * unable to obtain written informed consent from parent;
  * presence of congenital liver or renal, or metabolic diseases; and
  * ostomy caused by gastroschisis, omphalocele, imperforate anus, and perinatal asphyxia
  * unable to initiate enteral feeds after 28 days of ostomy placement.

Ages: 1 Day to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Average duration of exposure to PN (including Intralipid, IL) between the initial feeding and bowel reanastomosis | up to three years
  We hypothesize that the average duration of exposure to PN/IL of the infants receiving ML/FO will be less than that of infants receiving usual care. The ratio of enteral to parenteral nutrition in the infants receiving ML/FO will be greater than that of infants receiving usual care.

SECONDARY OUTCOMES:
Average weight gain (g/day)from initiating feeding to reanastomosis | up to three years
  We hypothesize that the average weight gain in infants receiving ML/FO will be greater than that of infants receiving usual care.
Average level of conjugated bilirubin and ostomy output of infants receiving ML/FO to the group receiving usual care between the initial feeding after placement of ostomy and reanastomosis | up to three years
  W hypothesize that the average level of conjugated bilirubin and ostomy output of infants receiving ML/FO will be less than that of infants receiving usual care.
Dietary fat and protein absorption, from initiating feeding to reanastomosis | up to three years
  Twenty-four hour stool (from ostomy) will be collected once per week after initiating feeding. Fecal fat and protein will be measured. Dietary fat and protein absorption will be calculated by subtracting fecal fat or protein from enteral dietary fat or protein, respectively.
  We hypothesize that infants receiving enteral ML/FO will have higher dietary fat and protein absorption than infants receiving routine care from initiating feeding to reanastomosis.
Expression of four key genes that play a crucial role in intestinal adaptation | up to four years
  RNA expression of four genes in small intestine, peptide YY (PYY), apical sodium dependent bile acid transport (ASBT), glucagon-like peptide-2 (GLP-2), and CD36 or fatty acid translocase (FAT), will be measured in both samples from stoma and distal mucous fistula sites.
Neurodevelopment outcomes and growth in the infants receiving ML/FO vs. in the infants receiving usual care at the 18-24 month of age. | up to 4.5 years
  We hypothesize that the early supplement of enteral ML/FO will have no adverse effect on the neurodevelopment outcomes and growth in the infants receiving ML/FO comparing to the infants receiving usual care at the 18-24 month of age.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Yang, MD, PhD, Principal Investigator — Wake Forest Univeristy Health Science
Locations (1):
- WFUHS Brenner Children's Hospital NICU, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Yang Q, Kock ND. Effects of dietary fish oil on intestinal adaptation in 20-day-old weanling rats after massive ileocecal resection. Pediatr Res. 2010 Sep;68(3):183-7. doi: 10.1203/PDR.0b013e3181eb2ee5. PMID 20531250
- [Background] Yang Q, Lan T, Chen Y, Dawson PA. Dietary fish oil increases fat absorption and fecal bile acid content without altering bile acid synthesis in 20-d-old weanling rats following massive ileocecal resection. Pediatr Res. 2012 Jul;72(1):38-42. doi: 10.1038/pr.2012.41. Epub 2012 Mar 23. PMID 22447320
- [Result] Yang Q, Welch CD, Ayers K, Turner C, Pranikoff T. Early enteral fat supplementation with microlipid(R) and fish oil in the treatment of two premature infants with short bowel. Neonatology. 2010;98(4):348-53. doi: 10.1159/000316067. Epub 2010 Oct 27. PMID 20980771
- [Result] Woods CW, Ayers K, Turner C, Pranikoff T and Yang Q. A Novel Nutritional Approach to Prevent Parenteral Nutrition-Associated Cholestasis in Two Premature Infants with Short Bowel Syndrome. ICAN: Infant, Child, & Adolescent Nutrition 2013 5: 32-36
- [Result] Yang Q, Ayers K, Chen Y, Helderman J, Welch CD, O'Shea TM. Early enteral fat supplement and fish oil increases fat absorption in the premature infant with an enterostomy. J Pediatr. 2013 Aug;163(2):429-34. doi: 10.1016/j.jpeds.2013.01.056. Epub 2013 Feb 28. PMID 23453547
- [Derived] Younge N, Yang Q, Seed PC. Enteral High Fat-Polyunsaturated Fatty Acid Blend Alters the Pathogen Composition of the Intestinal Microbiome in Premature Infants with an Enterostomy. J Pediatr. 2017 Feb;181:93-101.e6. doi: 10.1016/j.jpeds.2016.10.053. Epub 2016 Nov 15. PMID 27856001
- [Derived] Yang Q, Ayers K, Chen Y, O'Shea TM. Early enteral fat supplementation improves protein absorption in premature infants with an enterostomy. Neonatology. 2014;106(1):10-6. doi: 10.1159/000357554. Epub 2014 Mar 6. PMID 24603562